CLINICAL TRIAL: NCT04560595
Title: Remote Guided Caffeine Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00250925; R01DA003890 (NIH)
Record Dates: First submitted 2020-09-08; First posted 2020-09-23 (Actual); Results first posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Caffeine Dependence; Anxiety; Sleep Disturbance; Gastrointestinal Dysfunction; Sleep Initiation and Maintenance Disorders; Caffeine; Sleep Disorder; Caffeine; Caffeine-Induced Anxiety Disorder; Caffeine Withdrawal; Caffeine-Induced Sleep Disorder, Without Use Disorder; Caffeine Abuse; Insomnia; Anxiety Disorders; Sleep Disorder; Heartburn; Diarrhea
Keywords: caffeine; caffeine reduction; online study; manualized treatment; caffeine fading; remote intervention; remote trial
MeSH Terms: conditions — Anxiety Disorders; Parasomnias; Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders; Heartburn; Diarrhea

STUDY DESIGN:
Intervention Model Description: Caffeine consumption and secondary measures will be examined before, during, and after the caffeine reduction intervention and compared between immediate and delayed treatment groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caffeine Reduction Manual, Immediate Treatment Group (Experimental): Weekly caffeine consumption is to be measured before and after using the caffeine reduction program, which has been summarized in a "Guide to Caffeine Reduction and Cessation" manual to help people reduce their caffeine use. Those in the immediate treatment group will receive the guide immediately after screening.
  Interventions: Behavioral: Caffeine Reduction Manual
- Caffeine Reduction Manual, Delayed Treatment Group (Experimental): Weekly caffeine consumption is to be measured before and after using the caffeine reduction program, which has been summarized in a "Guide to Caffeine Reduction and Cessation" manual to help people reduce their caffeine use. Those in the delayed treatment group will receive the guide seven weeks after screening.
  Interventions: Behavioral: Caffeine Reduction Manual

INTERVENTIONS:
Behavioral: Caffeine Reduction Manual — We will provide participants with a Guide to Caffeine Reduction and Cessation in order to help the reduce their caffeine use and determine their ratings of treatment acceptability.
  Other Names: Johns Hopkins Guide to Caffeine Reduction and Cessation

SUMMARY:
The purpose of this online research study is to determine whether or not a gradual caffeine reduction program developed at Johns Hopkins can help people reduce their caffeine use. The investigators will provide materials to help guide caffeine reduction and ask questions to track caffeine use over several weeks. The investigators will also assess how reducing caffeine may benefit common caffeine-related problems such as anxiety, sleep disturbances, and gastrointestinal distress. The study will also determine whether or not people like participating in this caffeine reduction program in an online format.

DETAILED DESCRIPTION:
There is emerging evidence that some individuals have difficulty cutting down or eliminating caffeine consumption in spite of clinically significant problems exacerbated by caffeine use. This study will evaluate whether a caffeine reduction program developed at Johns Hopkins can help people reduce their caffeine use in an online format. Volunteers will participate in an intervention study conducted entirely online, including video visits for screening, instructions for caffeine reduction, and follow up. The study also involves filling out online surveys sent via email and text message. During screening, participants will be asked questions about their personal characteristics including demographic information, weekly caffeine consumption, and general medical history. Participants who are determined to be eligible after screening will be randomized to either the immediate or delayed treatment group. Those in the immediate treatment group will have their next session immediately after screening while those in the delayed treatment group will have their next session 7 weeks after screening. At this session, participants receive a digital copy of a caffeine reduction manual and instructions on how to gradually cut down caffeine. After this, participants will complete weekly online surveys over six weeks. Participants will complete two follow-up video visits at 7 and 14 weeks after participants received the caffeine reduction instructions. The investigators will measure caffeine consumption over time using the online surveys and interview questions during video visits, and the investigators will also measure how various caffeine related problems may improve during caffeine reduction, such as sleep problems, gastrointestinal issues, and anxiety. During the end of study sessions, participants will answer questions related to acceptability of the online format and report on participants' current caffeine use.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old
* Reside in the United States
* Read, write, and speak English fluently
* Able to access a video camera on a smart phone, tablet, or other computer
* Able to receive text messages or emails (or both)
* Suitable caffeine consumption
* Indicate suitable reason for caffeine reduction
* Interested in getting help to gradually reduce or eliminate caffeine consumption as part of a research study

Exclusion Criteria:

* Any current medical or psychiatric disorder or symptoms that, in the opinion of the investigators, may interfere with or preclude completion of the study [many psychiatric or medical concerns such as insomnia or anxiety are not anticipated to interfere with study participation and will not generally be exclusionary]

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dustin Lee, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Behavioral Pharmacology Research Unit, Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
There is not currently a plan to make individual participant data available to other researchers.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Caffeine Reduction Manual, Immediate Treatment Group | Caffeine Reduction Manual, Delayed Treatment Group
Started | 53 | 56
Completed | 48 | 45
Not Completed | 5 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Caffeine Reduction Manual, Immediate Treatment Group | Caffeine Reduction Manual, Delayed Treatment Group | Total
Number analyzed (Participants) | 53 | 56 | 109
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 53 | 56 | 109
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.36 (15.42) | 41.96 (14.14) | 43.61 (14.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 29 | 54
  Male | 28 | 27 | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 1 | 6
  Not Hispanic or Latino | 48 | 55 | 103
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 5 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 42 | 42 | 84
  More than one race | 3 | 6 | 9
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 53 | 56 | 109

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Retention as Assessed by Number of Participants With Completed Assessments
Description: To determine to what extent participants will engage with a remote caffeine reduction intervention for caffeine-related problems and find it acceptable, we will calculate the percentage of completed assessments for each video visit among eligible participants.
Time Frame: Treatment Visit, 7-Week Follow-Up, 14-Week Follow-Up
Population: All available data analyzed at each timepoint
Measure: Count of Participants; unit: Participants
Arm/Group | Caffeine Reduction Manual, Immediate Treatment Group | Caffeine Reduction Manual, Delayed Treatment Group
Number analyzed (Participants) | 53 | 56
Participants
  Treatment Visit | 51 | 51
  7-Week Follow-Up | 50 | 46
  14-Week Follow-Up | 48 | 45

2. Primary Outcome: Treatment Acceptability as Assessed by Treatment Acceptability Questionnaire
Description: At the 7 Weeks Follow-Up video visit, we will use an internally-developed standardized treatment acceptability questionnaire to determine self-reported agreement with two items on the treatment acceptability survey (i.e., "Overall, was the Guide to Caffeine Reduction and Cessation easy to use?", and "Overall, was the guide to Caffeine reduction and Cessation helpful?"). Each question is scored on a scale from 0-3, for a total score range of 0-6, where lower scores indicate less acceptability (e.g., 0=not at all easy, not at all helpful; 3 = very easy, very helpful).
Time Frame: 7 weeks Follow-Up visit
Population: Analysis population consists of participants who completed the week 7 end of treatment visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caffeine Reduction Manual, Immediate Treatment Group | Caffeine Reduction Manual, Delayed Treatment Group
Number analyzed (Participants) | 49 | 46
score on a scale | 2.50 (0.52) | 2.55 (0.50)

3. Secondary Outcome: Change in Caffeine Consumption (in Milligrams)
Description: To determine to what extent participants are successfully able to reduce their caffeine consumption following the remote intervention, we will assess caffeine consumption as determined by the standardized caffeine assessments at 7 week post-treatment follow-ups and compare this with consumption at the screening televisit. Based on participant responses to the number, type, and amount of caffeinated beverages, caffeine consumption is calculated at each assessment in milligrams (mg).
Time Frame: Baseline, Treatment Visit, 7-Week Follow-Up, 14-Week Follow-Up
Population: All available data analyzed at each timepoint
Measure: Mean (Standard Deviation); unit: milligrams of caffeine
Arm/Group | Caffeine Reduction Manual, Immediate Treatment Group | Caffeine Reduction Manual, Delayed Treatment Group
Number analyzed (Participants) | 53 | 56
milligrams of caffeine
  Baseline Visit | 617.34 (354.82) | 516.30 (218.79)
  Treatment Visit: number analyzed (Participants) | 51 | 51
  Treatment Visit | 602.90 (334.29) | 553.60 (246.62)
  7-Week Follow-Up: number analyzed (Participants) | 50 | 46
  7-Week Follow-Up | 221.58 (235.60) | 173.14 (161.72)
  14-Week Follow-Up: number analyzed (Participants) | 48 | 45
  14-Week Follow-Up | 219.61 (199.06) | 195.56 (207.39)

4. Secondary Outcome: Change in Caffeine-related Problems as Assessed by Past-7 Days Standardized Items
Description: To determine to what extent participants report improvement in common caffeine-related problems following the remote intervention, we have developed a standardized 19-Item Caffeine Use Disorder measure of the extent to which common problems related to excessive caffeine consumption bothered participants within the past 7 days, e.g., "During the past 7 days, I have consumed caffeine in larger amounts or over a longer period than I intended." Participants rate the extent to which these problems bothered them on a scale from 0-3 where 0 = not at all a problem and 3 = major problem. The total possible scale range is from 0-57 (because the scores of 0-3 are summed for the 19 items). Higher sum scores on the measure indicate greater caffeine-related problems.
Time Frame: Baseline, 7-Week Follow-Up, 14-Week Follow-Up
Population: All available data analyzed at each timepoint
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caffeine Reduction Manual, Immediate Treatment Group | Caffeine Reduction Manual, Delayed Treatment Group
Number analyzed (Participants) | 53 | 56
score on a scale
  Baseline | 17.85 (10.57) | 19.23 (10.88)
  7-Week Follow-Up: number analyzed (Participants) | 50 | 46
  7-Week Follow-Up | 5.52 (4.89) | 6.28 (5.92)
  14-Week Follow-Up: number analyzed (Participants) | 48 | 45
  14-Week Follow-Up | 4.26 (6.25) | 4.69 (5.53)

5. Secondary Outcome: Change in Anxiety as Assessed by the PROMIS-Anxiety-8a
Description: To determine whether caffeine reduction is accompanied by a reduction in day-to-day anxiety, we will utilize the Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety 8a assessment. The questionnaire asks the extent to which anxiety-related items affected the participants over the past 7 days on a scale of 1 (never) to 5 (always) with a total raw score range of 8-40 in which higher scores reflect greater anxiety. Raw scores are then translated into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. A higher PROMIS T-score represents more of the concept being measured. For negatively-worded concepts like anxiety, a T-score of 60 is one SD worse than average. By comparison, an anxiety T-score of 40 is one SD better than average. A score of less than 55 is none to slight, 55.0-59.9 is mild, 60.0-69.9 is moderate, and 70 and over is severe.
Time Frame: Baseline, 7-Week Follow-Up, 14-Week Follow-Up
Population: All available data analyzed at each timepoint
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Caffeine Reduction Manual, Immediate Treatment Group | Caffeine Reduction Manual, Delayed Treatment Group
Number analyzed (Participants) | 53 | 56
T-score
  Baseline | 57.31 (7.30) | 57.38 (5.96)
  7-Week Follow-Up: number analyzed (Participants) | 50 | 46
  7-Week Follow-Up | 49.78 (8.62) | 49.55 (7.44)
  14-Week Follow-Up: number analyzed (Participants) | 48 | 45
  14-Week Follow-Up | 49.82 (7.69) | 50.6 (8.78)

6. Secondary Outcome: Change in Anxiety as Assessed by the GAD-7
Description: To determine whether caffeine reduction is accompanied by a reduction in day-to-day anxiety, we will utilize the Generalized Anxiety Disorder-7 (GAD-7). The GAD-7 consists of items asking the participant to rate on a scale of 0 (not at all) to 3 (nearly every day) the extent they have experienced anxiety related symptoms. The scoring range is 0-21 and higher scores indicate greater anxiety related symptoms.
Time Frame: Baseline, 7-Week Follow-Up, 14-Week Follow-Up
Population: All available data analyzed at each timepoint
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caffeine Reduction Manual, Immediate Treatment Group | Caffeine Reduction Manual, Delayed Treatment Group
Number analyzed (Participants) | 53 | 56
score on a scale
  Baseline | 6.96 (5.79) | 6.13 (5.39)
  7-Week Follow-Up: number analyzed (Participants) | 50 | 46
  7-Week Follow-Up | 3.76 (4.84) | 3.13 (3.20)
  14-Week Follow-up: number analyzed (Participants) | 48 | 45
  14-Week Follow-up | 3.00 (4.34) | 3.24 (4.03)

7. Secondary Outcome: Change in Sleep Problems as Assessed by the PROMIS Sleep Disturbance 8a
Description: To determine whether caffeine reduction is accompanied by a reduction in sleep problems, we will utilize the PROMIS Sleep Disturbance 8a assessment. The questionnaire asks the extent to which sleep-related items affected the participants over the past 7 days on a scale of 1 (not at all) to 5 (very much). The raw scoring range is 8-40 and higher scores reflect greater sleep disturbance. Raw scores are then translated into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. A higher PROMIS T-score represents more of the concept being measured. For negatively-worded concepts like sleep disturbance, a T-score of 60 is one SD worse than average. By comparison, T-score of 40 is one SD better than average. A T-score of 50 or above is often considered a clinically significant level of sleep disturbance.
Time Frame: Baseline, 7-Week Follow-Up, 14-Week Follow-Up
Population: All available data analyzed at each timepoint
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Caffeine Reduction Manual, Immediate Treatment Group | Caffeine Reduction Manual, Delayed Treatment Group
Number analyzed (Participants) | 53 | 56
T-score
  Baseline | 55.54 (6.96) | 53.94 (6.57)
  7-Week Follow-Up: number analyzed (Participants) | 50 | 46
  7-Week Follow-Up | 47.09 (9.12) | 46.57 (6.74)
  14-Week Follow-Up: number analyzed (Participants) | 48 | 45
  14-Week Follow-Up | 45.13 (7.17) | 46.20 (6.56)

8. Secondary Outcome: Change in Sleep Problems as Assessed by the PSQI
Description: To determine whether caffeine reduction is accompanied by a reduction in sleep problems, we will utilize the Pittsburgh Sleep Quality Index (PSQI), which contains 19 self-rated items and 7 sub-scales for different components where a score of 0 indicates no difficulty and a score of 3 indicates severe difficulty. The scoring range is 0-21 and higher global scores indicate greater sleep difficulties.
Time Frame: Baseline, 7-Week Follow-Up, 14-Week Follow-Up
Population: All available data analyzed at each timepoint
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caffeine Reduction Manual, Immediate Treatment Group | Caffeine Reduction Manual, Delayed Treatment Group
Number analyzed (Participants) | 53 | 56
score on a scale
  Baseline | 9.21 (3.64) | 8.96 (3.16)
  7-Week Follow-Up: number analyzed (Participants) | 50 | 46
  7-Week Follow-Up | 6.80 (3.56) | 6.15 (2.97)
  14-Week Follow-Up: number analyzed (Participants) | 48 | 45
  14-Week Follow-Up | 5.60 (3.39) | 5.76 (2.80)

9. Secondary Outcome: Change in Gastrointestinal Problems as Assessed by the PROMIS Reflux-13a
Description: To determine whether caffeine reduction is accompanied by a reduction in gastrointestinal problems, we will utilize the PROMIS Reflux-13a. These items ask the extent to which gastrointestinal-related items affected the participants over the past 7 days on a scale of 1 (never) to 5 (always). The scoring range of raw scores is 13-65 and higher scores reflect greater gastrointestinal problems. Raw scores are then translated into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. A higher PROMIS T-score represents more of the concept being measured. For negatively-worded concepts like reflux, a T-score of 60 is one SD worse than average. By comparison, an anxiety T-score of 40 is one SD better than average.
Time Frame: Baseline, 7-Week Follow-Up, 14-Week Follow-Up
Population: All available data analyzed at each timepoint.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Caffeine Reduction Manual, Immediate Treatment Group | Caffeine Reduction Manual, Delayed Treatment Group
Number analyzed (Participants) | 53 | 56
T-score
  Baseline | 48.35 (8.71) | 49.32 (7.49)
  7-Week Follow-Up: number analyzed (Participants) | 50 | 46
  7-Week Follow-Up | 40.57 (7.17) | 40.73 (5.88)
  14-Week Follow-Up: number analyzed (Participants) | 48 | 45
  14-Week Follow-Up | 40.28 (7.32) | 40.73 (6.34)

10. Secondary Outcome: Change in Gastrointestinal Problems as Assessed by the GSRS
Description: To determine whether caffeine reduction is accompanied by a reduction in gastrointestinal problems, we will utilize the Gastrointestinal Symptoms Rating Scale (GSRS) which consists of 15 items describing gastrointestinal distress where responses range from 0 (no discomfort at all) to 6 (very severe discomfort). The scoring range is 0-90 and higher scores indicate more severe gastrointestinal symptoms.
Time Frame: Baseline, 7-Week Follow-Up, 14-Week Follow-Up
Population: All available data analyzed at each timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caffeine Reduction Manual, Immediate Treatment Group | Caffeine Reduction Manual, Delayed Treatment Group
Number analyzed (Participants) | 53 | 56
score on a scale
  Baseline | 16.11 (12.84) | 17.64 (15.60)
  7-Week Follow-Up: number analyzed (Participants) | 50 | 46
  7-Week Follow-Up | 8.08 (8.28) | 8.98 (8.86)
  14-Week Follow-Up: number analyzed (Participants) | 48 | 45
  14-Week Follow-Up | 6.96 (9.36) | 9.11 (9.11)

11. Secondary Outcome: Change in Gastrointestinal Problems as Assessed by the PROMIS Diarrhea-6a
Description: To determine whether caffeine reduction is accompanied by a reduction in gastrointestinal problems, we will utilize the PROMIS Diarrhea-6a. These items ask the extent to which gastrointestinal-related items affected the participants over the past 7 days on a scale of 1 (never) to 5 (always). The raw scoring range is 6-30 and higher scores reflect greater gastrointestinal problems. Raw scores are then translated into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. A higher PROMIS T-score represents more of the concept being measured. For negatively-worded concepts like diarrhea, a T-score of 60 is one SD worse than average. By comparison, an anxiety T-score of 40 is one SD better than average.
Time Frame: Baseline, 7-Week Follow-Up, 14-Week Follow-Up
Population: All available data analyzed at each timepoint.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Caffeine Reduction Manual, Immediate Treatment Group | Caffeine Reduction Manual, Delayed Treatment Group
Number analyzed (Participants) | 53 | 56
T-score
  Baseline | 51.31 (9.07) | 50.70 (8.81)
  7-Week Follow-Up: number analyzed (Participants) | 50 | 46
  7-Week Follow-Up | 43.55 (7.05) | 43.61 (5.92)
  14-Week Follow-Up: number analyzed (Participants) | 48 | 45
  14-Week Follow-Up | 44.35 (7.59) | 45.02 (6.91)

ADVERSE EVENTS:
Time Frame: Up to 14 weeks
Arm/Group | Caffeine Reduction Manual, Immediate Treatment Group | Caffeine Reduction Manual, Delayed Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/56
Other Adverse Events (participants affected / at risk) | 0/53 | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-07): https://cdn.clinicaltrials.gov/large-docs/95/NCT04560595/Prot_SAP_000.pdf